CLINICAL TRIAL: NCT06720597
Title: Utilizing EndoPAT Device for Endothelial Dysfunction Assessment in Erectile Dysfunction and Hormonal Therapy
Brief Title: EndoPAT Device for Endothelial Dysfunction in ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Faysal Yafi, Associate Professor of Urology Director of Men's Health and Newport Urology Chief, Division of Men's Health and Reconstructive Urology, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5526
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Erectile Dysfunction; Hypogonadism, Male; Endothelial Dysfunction
Keywords: EndoPAT; Erectile Dysfunction; Hypogonadism; Endothelial Dysfunction; ED; Testosterone
MeSH Terms: conditions — Erectile Dysfunction; Eunuchism; Hypogonadism

STUDY DESIGN:
Intervention Model Description: Study groups:
  1. Vasculogenic ED confirmed by penile Doppler ultrasound Population: 40 men aged 18 or above years diagnosed with vasculogenic ED Intervention: None. Assessments: Endothelial function will be assessed using the EndoPAT device at baseline, 3 months, and 6 months post-intervention.
  2. PDE5 Inhibitor Therapy in Men with Vasculogenic Erectile Dysfunction (ED) Population: 40 men aged 18 or above years diagnosed with vasculogenic ED. Intervention: Daily low-dose PDE5 inhibitor therapy. Assessments: Endothelial function will be assessed using the EndoPAT device at baseline, 3 months, and 6 months post-intervention.
  3. Testosterone Therapy in Hypogonadal Men Population: 40 hypogonadal men aged 18 or above Intervention: Testosterone therapy as per clinical guidelines. Assessments: Endothelial function will be assessed using the EndoPAT device at baseline, 3 months, and 6 months post-intervention.
Masking Description: The data analysis will be conducted by statisticians blinded to the intervention status to reduce analysis bias. Data coding will be used to ensure that statisticians are unaware of the group assignments during the analysis phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PDE5 Inhibitor Therapy in Men with Vasculogenic Erectile Dysfunction (ED) (Active Comparator): Population: 40 men aged 18 or above years diagnosed with vasculogenic ED. Intervention: Daily low-dose PDE5 inhibitor therapy. Assessments: Endothelial function will be assessed using the EndoPAT device at baseline, 3 months, and 6 months post-intervention.
  Interventions: Drug: Daily low-dose PDE5 inhibitor therapy
- Testosterone Therapy in Hypogonadal Men (Active Comparator): Population: 40 hypogonadal men aged 18 or above Intervention: Testosterone therapy as per clinical guidelines. Assessments: Endothelial function will be assessed using the EndoPAT device at baseline, 3 months, and 6 months post-intervention.
  Interventions: Drug: Testosterone therapy as per clinical guidelines.
- Vasculogenic ED confirmed by penile Doppler ultrasound (No Intervention): Population: 40 men aged 18 or above years diagnosed with vasculogenic ED. Intervention: None Assessments: Endothelial function will be assessed using the EndoPAT device at baseline, 3 months, and 6 months post-intervention.

INTERVENTIONS:
Drug: Daily low-dose PDE5 inhibitor therapy — Neither arm of the study includes a control group, and the two interventions will not be compared directly. The primary objective is to evaluate endothelial function using the EndoPAT device at baseline, 3 months, and 6 months following the intervention in each arm.
  Arms: PDE5 Inhibitor Therapy in Men with Vasculogenic Erectile Dysfunction (ED)
Drug: Testosterone therapy as per clinical guidelines. — Neither arm of the study includes a control group, and the two interventions will not be compared directly. The primary objective is to evaluate endothelial function using the EndoPAT device at baseline, 3 months, and 6 months following the intervention.
  Arms: Testosterone Therapy in Hypogonadal Men

SUMMARY:
To assess endothelial dysfunction in young men (aged 30-50) with vasculogenic ED identified through penile Doppler ultrasound.

To evaluate changes in endothelial function using EndoPAT before and 3-6 months after daily low-dose phosphodiesterase type 5 (PDE5) inhibitor therapy.

To investigate endothelial function alterations in hypogonadal patients before and 3-6 months after initiating testosterone (T) therapy

DETAILED DESCRIPTION:
Endothelial Dysfunction and Cardiovascular Health: Endothelial dysfunction is characterized by impaired endothelium-dependent vasodilation, which is a critical factor in the development and progression of cardiovascular diseases. The endothelium, the thin layer of cells lining blood vessels, plays a pivotal role in vascular health by regulating blood flow, coagulation, and immune function. When the endothelium is not functioning properly, it can lead to a range of cardiovascular conditions, including atherosclerosis, hypertension, and erectile dysfunction (ED).

Erectile Dysfunction and Endothelial Dysfunction: ED is often an early marker of endothelial dysfunction and cardiovascular diseases. Vasculogenic ED, in particular, is linked to poor endothelial health, where impaired blood flow to the penile tissue results in the inability to achieve or maintain an erection. This condition shares common risk factors with other cardiovascular diseases, such as diabetes, hypertension, and hyperlipidemia, highlighting the interconnected nature of endothelial health and ED.

Hormonal Therapy and Endothelial Function: Testosterone therapy (T therapy) is commonly used to treat hypogonadism in men, a condition characterized by low testosterone levels. Hypogonadism itself is associated with an increased risk of cardiovascular diseases, and testosterone therapy has been shown to have varying effects on endothelial function. While some studies suggest that testosterone may improve endothelial health, others indicate potential risks, necessitating further research to clarify its impact.

Current Gaps in Knowledge:

Prevalence of Endothelial Dysfunction in Young Men with ED: While the association between endothelial dysfunction and ED is established, there is a need for precise data on the prevalence and extent of endothelial dysfunction specifically in young men with vasculogenic ED. Understanding this prevalence can inform targeted treatment strategies.

Impact of PDE5 Inhibitors on Endothelial Function: Phosphodiesterase type 5 (PDE5) inhibitors are a first-line treatment for ED, known to improve erectile function by enhancing blood flow. However, their direct impact on endothelial function over time remains underexplored, particularly in terms of long-term cardiovascular outcomes.

Effects of Testosterone Therapy on Endothelial Health: The influence of testosterone therapy on endothelial function in hypogonadal men is not well understood. There is conflicting evidence on whether testosterone therapy confers cardiovascular benefits or risks, necessitating comprehensive studies to determine its effects.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 years old and above
* Diagnosed with erectile dysfunction or hypogonadism

Exclusion Criteria:

* Patients without the above criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Enrollment: 120 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Endothelial Function as Measured by Reactive Hyperemia Index (RHI) | At baseline, 3 months, and 6 months post-intervention
  Definition: RHI is a measure of endothelial function derived from the EndoPAT device, which assesses the endothelium's ability to respond to induced hyperemia.
  Measurement: RHI is calculated based on the changes in digital pulse volume during reactive hyperemia following a 5-minute arterial occlusion.
  Criteria for Evaluation:
  Baseline RHI: Measured before any intervention. Post-Intervention RHI: Measured at 3 months and 6 months post-intervention. Improvement in RHI: Defined as an increase in RHI scores from baseline to follow-up measurements.

SECONDARY OUTCOMES:
Cardiovascular Health Markers | From baseline to 3 months and 6 months post-intervention.
  Successful Outcome: Statistically significant improvements in blood pressure, lipid profile, and blood glucose levels from baseline to 3 and 6 months.
  Failure: No significant changes or worsening of cardiovascular health markers.
Sexual Function Scores | From baseline to 3 months and 6 months post-intervention.
  Successful Outcome: Statistically significant improvement in IIEF scores from baseline to 3 and 6 months.
  Failure: No significant changes or deterioration in sexual function scores.
Adverse Events | From baseline to 3 months and 6 months post-intervention.
  Successful Outcome: Minimal and non-severe adverse events reported. Failure: High frequency or severe adverse events necessitating discontinuation of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Faysal A Yafi, MD, Principal Investigator — University of California, Irvine
Locations (1):
- UCI Urology | Men's Health Center, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No